CLINICAL TRIAL: NCT06164639
Title: Investigation of Potential Biomarkers in Bronchoalveolar Lavage Fluid and Exploration of the Pathogenic Mechanism Via EIT Examination for Reflux Aspiration-induced Alveolar Injury.
Brief Title: Potential Biomarkers and Pathogenic Mechanism for Reflux Aspiration-induced Lung Injury.
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSICU20231130
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-12

CONDITIONS: ARDS, Human; Aspiration Pneumonia
Keywords: Aspiration Pneumonia; ARDS; cytokines; EIT
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — The collected bronchoalveolar lavage fluid contains cellular components. We will centrifuge and separate the cells and supernatant. The supernatant will be used to detect biomarkers, while the cells will be used for sequencing analysis to explore the underlying mechanisms for further study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Reflux aspiration group: Reflux aspiration group
  Interventions: Behavioral: aspiration; Diagnostic Test: bronchial alveolar fluid; Device: EIT V/Q test; Other: Nitric oxide inhalation
- Non-reflux aspiration group: Non-reflux aspiration group
  Interventions: Diagnostic Test: bronchial alveolar fluid

INTERVENTIONS:
Behavioral: aspiration — Based on whether the patient meets the diagnosis of aspiration pneumonia.
  Other Names: AP
  Groups: Reflux aspiration group
Diagnostic Test: bronchial alveolar fluid — Performing bronchoscopy.
  Other Names: BAL
Device: EIT V/Q test — Local pulmonary ventilation and perfusion are measured by electrical impedance tomography (EIT). For perfusion imaging, 10 ml of 5% saline is injected as a central venous bolus. The matching of ventilation and perfusion reveals intrapulmonary shunting.
  Groups: Reflux aspiration group
Other: Nitric oxide inhalation — According to the physician's judgment and the family members' consent, the patient is administered nitric oxide inhalation at a dosage of 20-30 parts per million (ppm).
  Groups: Reflux aspiration group

SUMMARY:
There is limited research on aspiration pneumonia-induced ARDS (Acute Respiratory Distress Syndrome), and currently there is a lack of studies on corresponding biomarkers and pathogenic mechanisms. We hypothesize that pH and amylase in BAL (Bronchoalveolar Lavage) may serve as candidate biomarkers for inhalation-induced ARDS. Furthermore, we use EIT analysis to explore the pathological mechanisms of ARDS induced by AP and evaluate the clinical value of NO in improving hypoxemia.

DETAILED DESCRIPTION:
Aspiration pneumonia leading to acute respiratory distress syndrome (ARDS) is not uncommon in clinical practice, but sometimes it occurs covertly and is not easily detected by doctors or family members. Sometimes, acute respiratory failure occurs suddenly due to massive aspiration. Aspiration of gastric contents is the main cause of reflux aspiration, and there is also aspiration of pharyngeal secretions in patients with impaired swallowing function. Finding the cause of ARDS is of great significance for guiding treatment and determining prognosis, but currently there is limited research on aspiration pneumonia leading to ARDS, and there is a lack of effective biomarkers in clinical practice. Fiberoptic bronchoscopy is a commonly used examination and treatment method for ARDS patients. We hypothesize that the detection of pH or amylase in bronchoalveolar lavage fluid (BALF) may have diagnostic significance for reflux aspiration-induced ARDS. Changes in cell subgroups and cytokines in BALF are important for understanding the pathogenesis. Therefore, in our prospective study, we collected BALF from patients admitted to the ICU who underwent endotracheal intubation due to ARDS and required bronchoscopy examination. We tested the pH and amylase levels in the lavage fluid. We analyzed the causes of ARDS and compared the differences in pH and amylase levels in BALF between patients with reflux aspiration-induced ARDS and non-reflux aspiration-induced ARDS. In addition, we will also explore the changes in cells, cytokines, and omics differences in BALF of confirmed cases of reflux aspiration-induced ARDS to search for possible pathogenic mechanisms. This study's use of bronchoscopy examination is in line with patient treatment needs and will not increase patient suffering or burden. Informed consent will be obtained from all patients admitted to the ICU with ARDS before enrollment.

Recently, a retrospective analysis comparing the differences in amylase and pancreatic enzyme levels in BALF between aspiration pneumonia and non-aspiration pneumonia was published in Pulmonology. Based on the number of cases and ROC results, PASS (2021, v21.0.3) was used, requiring 22 cases (11 each) with a 20% dropout rate, resulting in 28 cases (14 each). In statistical analysis, data is presented as mean ± standard deviation or the interquartile range (IQR) of 25-75% as the median. F test was performed to compare the means of the two groups. Student's t-test and Welch's t-test were used to compare values with and without homogeneity, respectively. One-way analysis of variance was used for multiple comparisons. Mann-Whitney U test and Wilcoxon signed-rank test were used for comparing median values between independent variables and dependent variables. Kruskal-Wallis test was used for multiple comparisons. Receiver operating characteristic (ROC) curve analysis was used to evaluate the clinical effectiveness of BAL-amylase and BAL-pH, and chi-square test was used to examine their relationship with risk factors for aspiration-induced ARDS. Univariate and multivariate logistic regression analyses were performed to investigate the relationship between BAL-amylase or BAL-pH and ARDS, expressed as odds ratios (OR) with 95% confidence intervals (CI). All analyses were conducted using PASS.

EIT is often used in ARDS patients to assess ventilation function and titrate appropriate PEEP. In these patients, we perform EIT for ventilation-perfusion detection as clinically needed. This is a non-invasive procedure, while blood gas analysis is also essential for ARDS detection. For some patients, when judged by doctors and consented by family members, we administer nitric oxide (NO) inhalation therapy, and conduct follow-up EIT after NO inhalation according to the patient's condition changes. Therefore, for patients with AP-ARDS, we also monitor the changes in EIT ventilation-perfusion and record the blood gas changes and CT findings.

ELIGIBILITY:
Inclusion Criteria:

The patient is between 18-99 years old. The patient meets the diagnostic criteria for ARDS upon admission to the ICU or during hospitalization, and requires mechanical ventilation with endotracheal intubation.

Within 24 hours of endotracheal intubation, bronchoscopy is performed for diagnostic or therapeutic purposes, and BALF is collected.

PH, amylase, and cytokines are tested within 24 hours. The patient, legal guardian, or authorized patient representative must voluntarily sign an informed consent form approved by the corresponding institutional review board. If the patient signs the consent form, the person obtaining consent must ensure that the patient is in a sufficient condition to provide informed consent.

Exclusion Criteria:

Clinical diagnosis of left ventricular failure Lung cancer-primary or metastatic Hematologic malignancy Acute gastrointestinal bleeding precluding enteral feeding Severe immunosuppression, defined as cytotoxic therapy within 15 days or White blood cell count of 5000 7) Use of steroids: 0.25 mg/kg/day of prednisone (or an equivalent dose of corticosteroids) Use of nonsteroidal anti-inflammatory (including aspirin) drugs within the last 24 hrs Known to be HIV positive Moribond at entry Pregnancy or positive pregnancy test

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS caused by inhalation pneumonia and patients with ARDS caused by other reasons.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
pepsin levels in BAL | Submit for examination within 24 hours after each BAL acquisition.
  Performing detection of pepsin in BAL

SECONDARY OUTCOMES:
PH levels in BAL | Submit for examination within 24 hours after each BAL acquisition.
  Performing detection of PH in BAL
EIT V/Q | Submit for examination within 30min after BAL acquisition.
  Local pulmonary ventilation and perfusion are measured by electrical impedance tomography (EIT). For perfusion imaging, 10 ml of 5% saline is injected as a central venous bolus. The matching of ventilation and perfusion reveals intrapulmonary shunting.
P/F ratio | All blood gas changes within 24 hours after enrollment
  Take the first blood gas after enrollment as the baseline, and record all blood gas values within 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No